CLINICAL TRIAL: NCT04803786
Title: Transition Experience of Persons With Narcolepsy Taking Oxybate in the Real-world (TENOR): A Patient-Centric, Prospective, Observational, Non-Interventional Study to Assess Dosing Regimen in Persons Switching From Xyrem to Xywav for the Treatment of Narcolepsy
Brief Title: A Patient-Centric, Prospective, Observational, Non-Interventional Switch Study of XYWAV in Narcolepsy
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: JZP258-402
Record Dates: First submitted 2021-03-09; First posted 2021-03-18 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transition from Xyrem to Xywav
  Interventions: Drug: Transition from Xyrem to Xywav

INTERVENTIONS:
Drug: Transition from Xyrem to Xywav — This is a single-group non-interventional study where participant's transitioning from Xyrem to Xywav will be observed. Investigational product (IP) or drug support or requested changes to their medication will not be provided to participants by Jazz Pharmaceuticals. The Xyrem and Xywav that the participants will take will be provided by the participant's health care provider.

SUMMARY:
The rationale for the patient-centric, prospective, observational, non-interventional study design of JZP258-402 is to evaluate the transition experience of participants with narcolepsy treated with oxybate and to examine the impact of transitioning from Xyrem to Xywav in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years or older
2. Diagnosis of type 1 or type 2 narcolepsy by a physician
3. Active prescription for Xyrem with a stable treatment regimen for at least 2 consecutive months
4. Transitioning from Xyrem to Xywav within the next or past 7 days (- 7 days or + 7 days from the first dose of Xywav)
5. Able to read and understand English
6. Able to access to a computer/smart phone with internet connection
7. Not currently a Jazz Pharmaceuticals employees or an immediate family member of a Jazz employee
8. Willing and able to comply with the study schedule
9. Willing and able to provide electronically written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female asges 18 years and older with diagnosis of type 1 or type 2 narcolepsy. On an active prescription for Xyrem with stable treatment for at least 2 consecutive months.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Increased/Decreased/Same Dose Transitioning from Xyrem to Xywav | Baseline to 21 Weeks
  • Difference between usual Xyrem total nightly dose and initial prescribed total nightly Xywav dose.

SECONDARY OUTCOMES:
Number Prescribed Dose Adjustments of Xywav | Baseline to 21 Weeks
  The number of dosing adjustments per participants and number of participants with one or more dosing adjustments during the Xywav Treatment Period (Period 2 to 5) by treating physician (dosing amount or number of nightly doses), details of adjustment, reason for adjustment and reason for unequal dosing will be summarized.
Duration of Time Between the Last Meal Relative to Dosing | Baseline to 21 Weeks
  Timing and type of last meal prior to the first dose will be collected using both Daily Diary and Weekly Lookback of Daily Diary. The timing will be collected as actual time (HH:MM) from Daily Diary and as categorical data of usual number of hours relative to first dose (<0.5 hours, ≥0.5 but <1 hours, ≥1 but <1.5 hours, ≥1.5 but <2 hours, ≥2 hours) from Weekly Lookback of Daily Diary. In order to evaluate the timing of last meal across all study periods, the Daily Diary entry will be converted into categorical data using the same value scale as Weekly Lookback of Daily Diary. The type of last meal prior to the first dose will be collected as categorical data (regular meal, snack, and beverage). For both timing and type of last meal prior to the first dose, the number of participants with each response will be summarized.

OTHER OUTCOMES:
Time to Achieve Stable Dose of Xywav | Baseline to 21 Weeks
  Stable dose is defined as the dose and regimen which remain unchanged for at least 2 weeks. Compliance is not considered in the derivation of the time to stable dose. The time to achieve stable dose will be summarized.
Number of Participants Achieving Treatment Adherence | Baseline to 21 Weeks
  Skipped doses will be collected using both the Daily Diary and Weekly Lookback Daily Diary. Skipped doses will be collected daily (yes/no) from the Daily Diary and as a weekly categorical variable (0, 1-2, 3-4, 5-6, or 7 days) from the Weekly Lookback of Daily Diary. In order to summarize skipped doses during the Xywav Treatment Period, the Daily Diary data will be converted to categorical data using the same categories as in the Weekly Lookback of Daily Diary. Skipped doses per week (0, 1-2, 3-4, 5-6, 7 days), most common dosing change (did not take Xywav, skipped first dose, skipped second dose, skipped third dose) and most common reasons for dosing change will be summarized.
Number of Participants Who Discontinued Xywav Administration | Baseline to 21 Weeks
  The number of participants who discontinued Xywav administration during the Xywav Treatment Period (Period 2 to 5).
Change in Short-term and Long-term Nausea Using Patient Global Impression of Change (PGI-C) | Baseline to 21 Weeks
  The PGI-C is a series of self-administered questions designed to measure the meaningfulness of change in symptoms following an intervention. The PGI-C is used to assess the change in excessive daytime sleepiness, cataplexy, and short- and long-term nausea since the transition from Xyrem to Xywav. It is a 7-point Likert-type rating scale from 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, to 7 = very much worse. The score is the sum of responses to each of the answer choices.
Changes in Sleep Pattern and Quality | Baseline to 21 Weeks
  Sleep pattern (how long usually took to fall asleep after the first dose, how long usually spent awake during the night) will be summarized. Sleep pattern and quality will be collected using both Daily Diary and Weekly Lookback of Daily Diary. The number of participants with each response to sleep quality (very poor ~ very good) and feeling on how rested/refreshed when woke-up for the day (not at all rested ~ very well rested) will be summarized by day and by week. In order to analyze the data together the intention is to combine the daily by deriving the categorical frequency for the responses so that it can be combined with the categorical data collected in the weekly diary. Which will allow for a full analysis of the change from the Baseline period (Xyrem) to Xywav Treatment Period (Period 2 to 5) will be summarized for weekly data collected during the Xywav Treatment Period (Period 2 to 5) using Weekly Lookback of Daily Diary.
Change in Epworth Sleepiness Scale (ESS) | Baseline to 21 Weeks
  The ESS is a self-administered questionnaire with 8 questions (Johns 1991, Johns 1992). Respondents rate on a 4-point scale (0-3) their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS total score (the sum of 8 item scores, 0-3) can range from 0 to 24. Higher ESS total scores are associated with higher sleep propensity in daily life, also referred to as 'daytime sleepiness'. The ESS has been validated in several conditions, including narcolepsy (Johns 1994).
Change in Functional Outcomes of Sleep Questionnaire (FOSQ-10) Total Score | Baseline to 21 Weeks
  The FOSQ-10 (Chasens 2009) is a self-administered questionnaire designed to assess the impact of daytime sleepiness on activities of daily living. It consists in 10 items measuring the participant's general productivity, activity level, vigilance, and intimacy and sexual relationships. For each item, participants are asked to rate the level of difficulty in completing an activity on a 4-point Likert scale, from 1 "Yes, extreme" to 4 "No"). From the FOSQ-10 a total score is calculated: a higher score indicates better functional status. The FOSQ-10 is a reduced version of the original FOSQ-30. The FOSQ-10 was tested and found to be a psychometrically strong instrument performing similarly to the long version.
Change in British Columbia Cognitive Complaint Inventory (BC-CCI) Total Score | Baseline to 21 Weeks
  The BC-CCI was developed to measure cognitive complaints in individuals with Major Depressive Disorder (MDD). It is a 6-item self-report measure that asks respondents to rate problems with specific cognitive symptoms over the past 7 days. A four point scale (0 "Not at all" to 3 "Very much") is used to rate each item. The total score (ranges from 0 to 18) that is generated assesses domains of memory, concentration, trouble expressing thoughts, word-finding, and problem solving. Higher scores indicate greater severity of cognitive impairment, with four established classification ranges for the BC-CCI total score: 0 to 4 = "broadly normal"; 5 to 8 = "mild" cognitive complaints; 9 to 14 = "moderate" cognitive complaints; and 15 to 18 = "severe" cognitive complaints. Three additional items that ask about how these symptoms impact work, relationships and social/recreational activities are also included to provide further information on the nature of functional impairment.
Change in Cataplexy using PGI-c | Baseline to 21 Weeks
  The PGI-C is a series of self-administered questions designed to measure the meaningfulness of change in symptoms following an intervention. The PGI-C is used to assess the change in excessive daytime sleepiness, cataplexy, and short- and long-term nausea since the transition from Xyrem to Xywav. It is a 7-point Likert-type rating scale from 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, to 7 = very much worse. The score is the sum of responses to each of the answer choices.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazz Pharmaceuticals Clinical Site, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No